CLINICAL TRIAL: NCT06181877
Title: The Effect Of Multifidus And Transversus Abdominis Muscle Activation Measured Under Ultrasound Guidance On Balance In Hemiplegic Patients
Brief Title: The Effect Of Multifidus And Transversus Abdominis Muscle Activation On Balance In Hemiplegic Patients
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nazlı Derya Bugdayci, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: ELMTRAMABHP
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Hemiplegia
Keywords: hemiplegia; transversus abdominis; multifidus; balance; stroke
MeSH Terms: conditions — Hemiplegia; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemiplegic Patients: Patients with hemiplegia after stroke

SUMMARY:
Patients with post-stroke hemiplegia may develop balance disorder and limitation in ambulation ability due to multiple mechanisms.

The effects of core muscles on maintaining normal posture, balance and ambulation ability are known. The positive effects of core stabilisation exercises on balance in hemiplegic patients have been shown in previous studies. In this study, we planned to investigate the effects of bilateral transversus abdominis and bilateral lumbar multifidus muscles on balance in patients with stroke-related hemiplegia.

DETAILED DESCRIPTION:
Loss of function in the trunk muscles of stroke patients leads to both balance problems and excessive effort to maintain balance. While ambulation ability of some patients is completely lost due to stroke, in others, impaired balance and increased postural oscillation lead to fear of falling and increased risk of falling.

In previous studies, it has been shown that there is a significant relationship between static balance and duration of hospital stay and functional abilities after stroke. In another study, it was shown that the control ability of the trunk muscles in the early post-stroke period was a strong factor affecting general life activities in the first six months after stroke.

Trunk muscles are innervated by both hemispheres unlike the extremities. Therefore, unilateral stroke may impair the function of trunk muscles on both the contralateral and ipsilateral sides. Several studies have shown dysfunction of bilateral trunk flexor, extensor and rotator muscles in patients with unilateral stroke.

Many studies have proven that core stabilisation exercises are effective on both balance and gait function and general life activities in hemiplegic patients.

The aim of this cross-sectional study was to investigate the effect of ultrasound-guided bilateral transversus abdominis and bilateral lumbar multifidus muscle activations on balance in hemiplegic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years
* Time after stroke must be at least 1 month
* Unilateral stroke
* Must be cognitively compatible in terms of cooperation
* Standing balance with/without support and/or sitting balance without support
* BMI<30

Exclusion Criteria:

* Patients with a history of hemiplegia in the opposite half of the body
* Patients with extruded or sequestered lumbar hernia and/or history of lumbar operation
* Patients with a history of lumbar vertebral fracture
* Patients with traumatic brain injury
* Patients with neuromuscular muscle disease that may lead to muscle atrophy
* Patients with sensory defects
* Patients with cerebellar defects
* Patients with vestibular balance disorders (vertigo, etc.)
* Patients with Parkinson's disease
* Patients with balance problems due to visual impairment
* Patients with pre-stroke balance problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 36 hemiplegic patients who met the inclusion criteria and did not meet the exclusion criteria
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | Same day with ultrasound-guided muscle measurement
  Patients' balance was evaluated using the Berg Balance Scale.
Postural Assessment Scale For Stroke Patients (PASS) | Same day with ultrasound-guided muscle measurement
  Posture change and posture maintenance scores of the patients were evaluated using PASS.
Functional Ambulation Category (FAC) | Same day with ultrasound-guided muscle measurement
  Ambulation ability of the patients was evaluated using FAC.

SECONDARY OUTCOMES:
Brunnstrom Stages | Same day with ultrasound-guided muscle measurement
  Limb function of the patients was evaluated using Brunnstrom Staging.
Transversus Abdominis Muscle Activation | BBS, PASS, FAC and Brunnstrom stages were measured immediately after recording.
  [(transversus abdominis contraction thickness)-(transversus abdominis resting thickness)]/transversus abdominis resting thickness
Multifidus Muscle Activation | BBS, PASS, FAC and Brunnstrom stages were measured immediately after recording.
  [(multifidus contraction thickness)-(multifidus resting thickness)]/multifidus resting thickness

CONTACTS AND LOCATIONS:
Overall Officials: NAZLI DERYA BUGDAYCI, MD, Principal Investigator — Istanbul Physical Therapy Rehabilitation Training & Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training & Research Hospital, Istanbul, Turkey (Türkiye)